CLINICAL TRIAL: NCT04792905
Title: Étude Exploratoire Des Performances de Diagnostic Électrocardiographique de l'Apple Watch augmentée d'un Algorithme d'Intelligence Artificielle
Brief Title: Exploratory Study of Apple Watch Electrocardiographic Diagnostic Performance Enhanced by an Artificial Intelligence Algorithm
Status: Completed | Type: Observational
Sponsor: Cardiologs Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: AI Watch
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Cardiologs — Two Apple Watch recordings (one recording with the watch on the wrist and one on the left side of the abdomen) interpreted by Cardiologs AI done simultaneously with each 12-lead ECG
  Other Names: Apple Watch

SUMMARY:
This observational exploratory prospective study will evaluate the performance on an Artificial Intelligence (AI) solution interpreting ECG (electrocardiogram) collected from an Apple Watch (AI-AW) in the detection of Atrial Fibrillation (AF)

DETAILED DESCRIPTION:
After being informed about the study, participants hospitalized for ablation or cardioversion or having a cardiac rhythm consultation at the investigational center will have Apple Watch ECG recordings done simultaneously with 12-lead ECG measurements performed in accordance with the existing in-stay subject monitoring protocol. AI-AW will be compared to standard manual 12-lead ECG reviewed by cardiologists for AF detection.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 22 or older, able and willing to participate in the study
* Patient admitted to hospital for ablation, cardioversion or cardiac electrophysiological exploration or who come for regular rhythmology consultations
* Patient who has read the information note and has given his or her consent before any procedure related to the study
* Patient affiliated to social security

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient with a pacemaker, implantable defibrillator or cardiac resynchronisation therapy device.
* Subject related to the investigator or any other staff member directly involved in the conduct of the study
* Patient incapable of giving consent, minor or adult patient protected by law

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 participants: patients hospitalized for ablation or cardioversion or patients having cardiac rhythm consultation and who have expressed non-opposition to participate to the study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Performance of AF detection | 1 day
  Performance of AF detection by an artificial intelligence (AI) solution interpreting ECG collected via Apple Watches (AI-AW), compared to physician's diagnosis from the 12 leads ECG

SECONDARY OUTCOMES:
AW versus AI-AW | 1 day
  Comparison of Apple Watch (AW) and AI-AW AF detection performance
AI-AW versus AI-12lead | 1 day
  Comparison of the performance of AF detection by AI-AW and AI applied to the 12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Fiorina, Dr, Principal Investigator — Institut Cardiologique Paris Sud Hôpital Privé Jacques Cartier
Locations (1):
- Institut Cardiologique Paris Sud Hôpital Privé Jacques Cartier, Massy, France

IPD SHARING:
Plan to Share IPD: No